CLINICAL TRIAL: NCT02297542
Title: Immune Response to High-Dose vs. Standard Dose Influenza Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Health Sciences North Research Institute (Other)
Collaborators: UConn Health (Other)
Responsible Party: Principal Investigator, Janet McElhaney, Senior Scientist, AMRIC, Professor (NOSM), Medical Lead for Senior's Care and Consulting Geriatrician (HSN), HSN Volunteer Association Chair in Geriatric Research, Health Sciences North Research Institute
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: NIH R01
Record Dates: First submitted 2014-11-03; First posted 2014-11-21 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-02

CONDITIONS: Elderly Immune System
Keywords: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flu Vaccine SD (Active Comparator): Fluzone Standard Dose Influenza Vaccine
  Interventions: Biological: Flu Vaccine
- Flu Vaccine HD (Active Comparator): Fluzone High Dose Influenza Vaccine
  Interventions: Biological: Flu Vaccine

INTERVENTIONS:
Biological: Flu Vaccine
  Other Names: Fluzone HD

SUMMARY:
This 5-year proposal is a randomized study of split-virus influenza vaccine (SVV) in a high-dose (HD) vs. standard-dose (SD) formulation in each of five influenza seasons to define the key determinants of vaccine-mediated protection against influenza and how these immunologic mediators may be enhanced by vaccination with a newly approved high-dose influenza vaccine in older people

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by the participant
2. Age 20-40 years old with no underlying chronic diseases or age ≥65 years old
3. Willing to receive influenza vaccination
4. Older cohort has received their influenza vaccine for the previous influenza season

   -

Exclusion Criteria:

1. Immunosuppressive disorders or medications (including oral prednisone in doses >10 mg daily)
2. Have not received influenza vaccination in the past or cannot be vaccinated due to previous severe reaction to influenza vaccine, egg, latex, or thimerosol allergies, or refusal of vaccination
3. Participant has received a community available influenza vaccine for the approaching influenza season
4. Females who are pregnant at Visit 1 (a pregnancy test will be administered for all females of child-bearing potential)

   -

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of Influenza Cases | five years
  Influenza surveillance includes weekly contact with study subjects to assess for any flu-like symptoms or acute respiratory infection (ARI), and include nasopharyngeal swabs (within 5 days of onset of symptoms) for polymerase chain reaction (PCR) detection of influenza virus and post-influenza season detection of an antibody response to influenza infection. Routine screen for symptoms of ARI will also occur at the 4, 10 and 20 week visits when blood samples are collected. Influenza illness will be documented by PCR detection of influenza during an IARI or seroconversion (4-fold rise in antibody titers) in association with an ARI. ARI includes upper (coryza or sore throat) or lower (cough or shortness of breath) respiratory tract symptoms, or headache, malaise, myalgia or fever (> 99°F or 37.3°C orally or 100°F rectally) [41]. as physician visits, hospitalizations and deaths attributed to acute cardiopulmonary illness and will be tracked through the influenza season.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E McElhaney, MD, Principal Investigator — Health Sciences North Research Institute
Locations (2):
- Center on Aging, UConn Health, Farmington, Connecticut, United States
- Health Sciences North Research Institute, Greater Sudbury, Ontario, Canada

REFERENCES:
- [Derived] McElhaney JE, Verschoor CP, Haynes L, Pawelec G, Loeb M, Andrew MK, Kuchel GA. Key Determinants of Cell-Mediated Immune Responses: A Randomized Trial of High Dose Vs. Standard Dose Split-Virus Influenza Vaccine in Older Adults. Front Aging. 2021 May;2:649110. doi: 10.3389/fragi.2021.649110. Epub 2021 May 21. PMID 35128529